CLINICAL TRIAL: NCT04667273
Title: Effectiveness of Neuromuscular Electrical Stimulation in Patients With Subacromial Impingement Syndrome: Randomized Controlled Study
Brief Title: Effectiveness of Neuromuscular Electrical Stimulation in Patients With Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ebru Kaya Mutlu, PT, Associate Prof. Dr, PhD, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/11
Record Dates: First submitted 2020-12-11; First posted 2020-12-14 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Shoulder impingement syndrome; Visual Analog Scale; Range of motion; Muscle strength; Sleep
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The sample of the study will consist of patients with subacromial impingement syndrome (SIS) who were referred to Istanbul University Cerrahpaşa Physical Therapy and Rehabilitation Department by an orthopedist. Forty eight SIS patients will be included in the study. Patients who meet the inclusion criteria will be divided into two groups.
  Group 1: Exercise Training+ Neuromuscular Electrical Stimulation Group 2: Exercise Training
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Training (ET) + Neuromuscular Electrical Stimulation (NMES) group (Experimental): volunteer patients with Subacromial Impingement Syndrome
  Interventions: Procedure: Neuromuscular Electrical Stimulation (NMES); Procedure: Exercise Training (ET)
- Exercise Training (ET) group (Other): volunteer patients with Subacromial Impingement Syndrome
  Interventions: Procedure: Exercise Training (ET)

INTERVENTIONS:
Procedure: Neuromuscular Electrical Stimulation (NMES) — In Neuromuscular Electrical Stimulation (NMES) application, 4 surface electrodes will be placed in the swollen part of the lower trapezius and serratus anterior muscles of each patient.
  NMES will be applied for 20 minutes in rehabilitation mode with a 4-channel device.
  Frequency: 80 Hz Amplitude: 0-100 mA (0-0.01 V) Current time-Pulse: 200 μsec Wave form: Biphasic Cycle time: 8 seconds of tetanic muscle stimulation for all patients, with a 2 second rise and fall time and stimulation It will be set as 3 seconds between. It is important to visually observe the contraction to determine the intensity of stimulation.
  Arms: Exercise Training (ET) + Neuromuscular Electrical Stimulation (NMES) group
Procedure: Exercise Training (ET) — Patients will do Wand exercises under the supervision of a physiotherapist. Wand exercises will include shoulder flexion, external rotation and abduction in the scaption position. In the first and second week, these exercises will be performed on the back, and from the third week on standing exercises.
  Exercises with the Theraband will be done in 3 sets, each set will consist of 10 repetitions. There will be a 1 minute rest period between sets. When the three sets are easily completed and there is no reported fatigue by the patient, the resistance will be increased by moving from yellow to red, from red to green, respectively, after 4 weeks.
  *For shoulder external rotators and serratus anterior muscles are strengthened without weight for the first 2 weeks, then 0.5 kg of dumbbells, in the supine position.
  While standing, the lower trapezius, upper trapezius and shoulder external rotators will be strengthened with theraband.

SUMMARY:
Subacromial Impingement Syndrome (SIS) is one of the musculoskeletal system problems. SIS, which is the most common cause of shoulder pain, constitutes 44-65% of complaints of shoulder pain. Studies have shown that exercise is effective in treating patients with SIS, but the effectiveness and superiority of Neuromuscular Electrical Stimulation (NMES) to each other is uncertain. NMES is widely applied in physiotherapy. In the SIS, the lower trapezius and serratus anterior muscle are affected. Therefore, our aim is to determine the effects of exercises and NMES used in patients with SIS on pain, range of motion (ROM), muscle strength and functional status, neck pain and sleep quality.

DETAILED DESCRIPTION:
The aim of this study investigate exercise training (ET) and ET combined with Neuromuscular Electrical Stimulation (NMES) on pain, range of motion (ROM), functional capacity, neck pain, sleep quality. The study will be included 48 volunteers with Subacromial Impingement Syndrome (SIS). The study's inclusion criteria are as follows: Having a diagnosis of subacute / chronic extrinsic SIS, 18 to 65 years of age and being volunteer. The exclusion criteria are as follows: Fracture or surgical history in the shoulder region, another diagnosis that can affect shoulder function, having received local corticosteroid injection / treatment in the shoulder joint within the last 3 months, neuromuscular disease, pregnancy, cancer, unstabil angina, communication problems, systemic inflammatory joint disease, situations where electrical stimulation and exercise are contraindicated, orthopedic, rheumatologic or congenital disease of the affected upper extremity. The sociodemographic data of the patients will be questioned. ET will be applied daily and NMES will be applied 2 days a week for 8 weeks. In addition, both groups will apply these exercises as a home program 3 times a day, 10 repetitions of each exercise. Pain intensity with Visual Analog Scale (VAS), range of motion (ROM) with goniometer, muscle strength with Hand-held Dynamometer, upper extremity function evaluation with Quick Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire, disability of neck level with Neck Disability Index, sleep quality with Pittsburgh Sleep Quality Index will be evaluated before and after treatment. All parameters will be compared between ET and ET+NMES group.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of subacute / chronic extrinsic SIS
* 18 to 65 years of age
* Being volunteer

Exclusion Criteria:

* Fracture or surgical history in the shoulder region
* Another diagnosis that can affect shoulder function
* Having received local corticosteroid injection / treatment in the shoulder joint within the last 3 months
* Neuromuscular disease
* Pregnancy
* Cancer
* Unstabil angina
* Communication problems
* Systemic inflammatory joint disease
* Situations where electrical stimulation and exercise are contraindicated
* Orthopedic, rheumatologic or congenital disease of the affected upper extremity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Disability Arm Shoulder Hand Questionnaire (DASH) | 8 weeks
  The DASH questionnaire is a region-specific, self-report scale to evaluate health status of upper extremity disabilities.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 8 weeks
  The VAS is used for which a patient is asked to indicate his/her perceived pain during the rest, activity and night times. Respondents will mark the location on the 10-centimeter (cm) line corresponding to the amount of pain they experienced.
Goniometer | 8 weeks
  Shoulder flexion, abduction, internal rotation, and external rotation, ROM will be measured by a universal goniometer.
Digital hand-held dynamometer | 8 weeks
  Shoulder flexion, extension, abduction, adduction, internal and external muscle strength measurements will be evaluated with a digital hand-held dynamometer called "Lafayette-Manual Muscle Tester". Before taking measurements, a few trials will be made by informing. Then the individual will be positioned according to the muscle to be tested, the device will be placed in the appropriate area of the muscle whose strength is to be measured, and the individual will be asked to maintain the specified position for each muscle. The evaluation is repeated twice and the value when the position starts to deteriorate will be recorded in newton as the result measurement.
Neck Disability Index | 8 weeks
  Pain related disability will be evaluated using the Turkish version of the Neck Disability Index. This questionnaire consists of 10 questions, each scored between 0 and 5. The final score of the questionnaire is obtained by adding the scores from each question. Disability levels of the patients are as follows: "no disability" (0-4), "mild disability" (5 14), "moderate disability" (15-24), "severe disability" (25 -34) and "complete disability".
Pittsburgh Sleep Quality Scale | 8 weeks
  The Pittsburgh Sleep Quality Scale will be applied to evaluate the sleep quality of the patients. With this scale, both the sleep quality of the patient is evaluated and whether there is a problem with daytime sleepiness is reviewed. In this evaluation; Subjective sleep quality, time to fall asleep, sleep duration, sleep quality, conditions that affect sleep, sleep substance use and daytime sleepiness are evaluated. Each area of the scale is calculated with scores ranging from 0 to 3, high scores indicate poor sleep quality. The total value in this test is a score between 0-21. Its Turkish validity and reliability were made in 1996 by Ağargün et al.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Kaya Mutlu, Assoc. Prof., Principal Investigator — İstanbul Üniversitesi- Cerrahpaşa İstanbul, Türkiye
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Bdaiwi AH, Mackenzie TA, Herrington L, Horsley I, Cools AM. Acromiohumeral Distance During Neuromuscular Electrical Stimulation of the Lower Trapezius and Serratus Anterior Muscles in Healthy Participants. J Athl Train. 2015 Jul;50(7):713-8. doi: 10.4085/1062-6050-50.4.03. Epub 2015 May 1. PMID 25933249
- [Result] Camargo PR, Alburquerque-Sendin F, Avila MA, Haik MN, Vieira A, Salvini TF. Effects of Stretching and Strengthening Exercises, With and Without Manual Therapy, on Scapular Kinematics, Function, and Pain in Individuals With Shoulder Impingement: A Randomized Controlled Trial. J Orthop Sports Phys Ther. 2015 Dec;45(12):984-97. doi: 10.2519/jospt.2015.5939. Epub 2015 Oct 15. PMID 26471852